CLINICAL TRIAL: NCT02640209
Title: Pilot Trial of Autologous T Cells Engineered to Express Anti-CD19 Chimeric Antigen Receptor (CART19) in Combination With Ibrutinib in Patients With Relapsed or Refractory CD19+ CLL or SLL
Brief Title: Pilot Trial Of Autologous T Cells Engineered To Express Anti-CD19 Chimeric Antigen Receptor (CART19)In Combination With Ibrutinib In Patients With Relapsed Or Refractory CD19+ Chronic Lymphocytic Leukemia (CLL)Or Small Lymphocytic Lymphoma (SLL)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study is terminated due to administrative reasons.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 18415, 823584
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2020-05

CONDITIONS: LYMPHOCYTIC LEUKEMIA (CLL) OR SMALL LYMPHOCYTIC LYMPHOMA (SLL)
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: CART 19

INTERVENTIONS:
Biological: CART 19 — The target dose range administered in this study is 1-5x108 CART-19 cells administered via split dosing: 10% on Day 1 (1-5x107 CART19), 30% on Day 1 (3x107-1.5x108 CART19), 60% on Day 2 (6x107-3x108 CART19).

SUMMARY:
Open-label pilot study to determine safety and efficacy of CART-19 cells in combination with ibrutinib. The target dose will be 1-5x10xE8 CART-19 transduced cells administered via split dosing: 10% on Day 1, 30% on Day 2, 60% on Day 3. 15 evaluable subjects (adults) with relapsed or refractory CLL/SLL who have achieved partial response or stable disease on ibrutinib therapy will be eligible to receive CART-19 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented CD19+ CLL or SLL
* Successful test expansion -cells (as described in Section 6.1)
* Patients must have failed at least 1 prior regimen before Ibrutinib (not including single agent rituximab or single agent corticosteroids)

  a. Note: Any relapse after prior autologous SCT will make the patient eligible regardless of other prior therapy.
* Patients must be currently receiving ibrutinib for at least 6 months prior to enrollment in the study and:

  1. Not experiencing any ≥ grade 2 non-hematologic ibrutinib-related toxicity
  2. The best response to ibrutinib therapy must not have exceeded partial response or stable disease (i.e. no CR or CRi)
  3. Note: Patients carrying a deletion at chromosome 17p (i.e. del[17p]), and/or TP53, BTK, and at the PLCγ2 loci mutations, will be eligible if they are receiving frontline therapy with ibrutinib.
* ECOG Performance status 0 or 1
* 18 years of age and older
* Adequate organ system function including:

  1. Creatinine < 1.6 mg/dl
  2. ALT/AST < 3x upper limit of normal
  3. Total Bilirubin <2.0 mg/dl with the exception of patients with Gilbert syndrome; patients with Gilbert syndrome may be included if their total bilirubin is ≥ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN.
* Patients with relapsed disease after prior allogeneic SCT (myeloablative or nonmyeloablative) will be eligible if they meet all other inclusion criteria and:

  1. Have no active GVHD and require no immunosuppression
  2. Are more than 6 months from transplant
* No contraindications for leukapheresis
* Left Ventricular Ejection fraction >40%
* Gives voluntary informed consent
* Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

* CLL patients with known or suspected transformed disease (i.e. Richter's transformation). Note: biopsy proven absence of transformation is not required.
* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* Patients with active CNS involvement with malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification.
* Subjects with clinically apparent arrhythmia or arrhythmias who are not stable on medical management within two weeks of enrollment.
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Saar Gill, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gill S, Vides V, Frey NV, Hexner EO, Metzger S, O'Brien M, Hwang WT, Brogdon JL, Davis MM, Fraietta JA, Gaymon AL, Gladney WL, Lacey SF, Lamontagne A, Mato AR, Maus MV, Melenhorst JJ, Pequignot E, Ruella M, Shestov M, Byrd JC, Schuster SJ, Siegel DL, Levine BL, June CH, Porter DL. Anti-CD19 CAR T cells in combination with ibrutinib for the treatment of chronic lymphocytic leukemia. Blood Adv. 2022 Nov 8;6(21):5774-5785. doi: 10.1182/bloodadvances.2022007317. PMID 35349631
- [Derived] Frey NV, Gill S, Hexner EO, Schuster S, Nasta S, Loren A, Svoboda J, Stadtmauer E, Landsburg DJ, Mato A, Levine BL, Lacey SF, Melenhorst JJ, Veloso E, Gaymon A, Pequignot E, Shan X, Hwang WT, June CH, Porter DL. Long-Term Outcomes From a Randomized Dose Optimization Study of Chimeric Antigen Receptor Modified T Cells in Relapsed Chronic Lymphocytic Leukemia. J Clin Oncol. 2020 Sep 1;38(25):2862-2871. doi: 10.1200/JCO.19.03237. Epub 2020 Apr 16. PMID 32298202